CLINICAL TRIAL: NCT01565759
Title: Investigation of the Effects of in Vivo Lithium Treatment on Gene Expression Levels Using Lymphoblastoid Cell Lines From Human Healthy Subjects
Brief Title: In Vivo Lithium Treatment Effects on Gene Expression Levels in Lymphoblastoid Cell Lines From Human Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CDHA-RS-2012-317; LithiumHV2012 (Registry Identifier: Manchia)
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Drug Mechanism
Keywords: Gene expression; Lithium; Healthy volunteers; Lymphoblastoid cell lines
MeSH Terms: interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lithium (Experimental): This will be a short-term longitudinal study of 4 weeks of duration. Twenty (20) healthy male subjects will be recruited and treated with lithium carbonate for 4 weeks. Lithium carbonate (150 mg, 300 mg, 600 mg) will be administered to the recruited subjects. The study will be performed in one centre at Capital District Health Authority - Dalhousie University, Halifax, Nova Scotia, Canada. Lithium serum levels will be tested at day 8, at day 14 and at the end of the treatment. Additional tests may be performed as necessary (as in the case of side effects).
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — The dose has been selected in order to achieve a therapeutic range of 0.6 - 0.8 mmol/L.
  Dose titration Day 1: 1 capsule of 300 mg at bedtime Days 2 to 7: 1 capsule of 600 mg at bedtime Day 8: lithium serum levels will be tested and the dose will be adjusted proportionally to a target range of 0.6 - 0.8 mmol/L by increments of 150 mg or 300 mg.

SUMMARY:
Psychiatric disorders often result from dysregulation in cellular and molecular mechanisms at the level of the brain. Unable to directly study brain tissues in patients affected by psychiatric conditions, researchers have created alternative experimental models that use different and easy to collect tissues. The underlying assumption is that by studying these "proxy" tissues, it is possible to obtain information on biological mechanisms that is a good approximation of what would be detected in the brain. One of the most established experimental models are lymphoblastoid cell lines derived from B-lymphocytes. Lymphocytes are present in the peripheral blood and can be easily collected and stored virtually forever after undergoing a special laboratory procedure that immortalize them. These cell lines have proved to be very useful in genetic and pharmacogenetic research and, using these, the investigators want to investigate the cellular effects of a mood stabilizing drug called lithium on this specific procedure that makes them virtually immortal. Two main reasons lead us to study this drug: 1) it is the most effective treatment in bipolar disorder, where approximately 30% of patients achieve complete illness remission with prevention of episode recurrence; 2) it has well established regulatory effects on the expression of specific target genes and proteins. The investigators can take advantage of these well-established properties of lithium in regulating the expression of genes, proteins, and enzymes in a stable manner. Conversely, these biological measures could be used as markers for the effects of lithium on the gene expression.

The purpose of this study is to learn more about the changes in the activity of genes in cells sampled from healthy individuals treated with lithium. By studying these cellular changes, the investigators hope to understand if lymphoblastoid cell lines are valid tools in psychiatric genetics research. Specifically, the investigators want to see how specially treated lymphoblastoid cell lines are influenced by external conditions and specifically lithium treatment at the moment of sampling. To do so, the investigators will measure the gene expression (i.e. how much gene is in the cell) of lymphoblastoid cell lines and compare the levels between those sampled before and after one month of lithium treatment.

DETAILED DESCRIPTION:
Background

One of the major limitations of psychiatric research is the necessity to use indirect methods to study neuronal functions. Among these, studies of transformed lymphocytes are an invaluable tool. Epstein Barr virus (EBV) transformed lymphoblasts can be used for a variety of purposes including in vitro studies of gene expression and investigations of cellular responses to pharmacological treatment. They can be kept and re-grown as needed and can often serve as a backup supply for DNA for genetic analyses. For these reasons, lymphoblasts cell lines (LCLs) have been collected and used by a number of research groups, including our own.

Most investigators work with the implicit assumption that such transformed cells represent trait characteristics of the person and their illness. In other words, the cell transformation and repeated passages are assumed to reduce the impact of any confounding factors present at the time of blood sampling and lymphocyte isolation. These factors may include, among others, the clinical state, the actual treatment, or time of the day. Surprisingly, we could not find any published data supporting or contradicting this assumption.

Here we propose to investigate the effects of one particular factor that may influence various cellular measures, namely in vivo drug treatment. Specifically, we are interested in assessing the effect of treatment with lithium, an ion that possesses mood-stabilizing properties. Indeed, lithium is the most effective treatment in bipolar disorder, with approximately 30% of patients achieving complete illness remission and prevention of episode recurrence (Baldessarini and Tondo, 2000; Garnham et al., 2007).

Rationale

Lithium has well established regulatory effects on the expression of specific target genes. Gene expression studies on LCLs from patients characterized for response to lithium treatment have identified a series of molecular target directly modulated by this drug. A microarray study (Sun et al., 2004) on LCLs of patients with BD characterized for full response to lithium demonstrated its effect in decreasing the expression of seven genes: somatostatin receptor type 2 (SSTR2), nuclear factor kappa-B DNA binding subunit (NF-kB), alpha1B-adrenoceptor (1B-AR), acetylcholine receptor protein alpha chain precursor (ACHR), cAMP-dependent 3', 5'-cyclic phosphodiesterase 4D (PDE4D), substance-P receptor (SPR), and ras-related protein (RAB7), the latter five being validated by Northern blotting analysis. Recently, using LCLs from three healthy subjects, Sugawara and coworkers (2010) identified 44 genes whose expression was regulated by lithium. Among the ten genes most down-regulated by lithium were Bax, zuotin related factor 1 (ZRF1) and thioredoxin domain containing 13 (TXNDC13), while platelet-activating factor acetylhydrolase, isoform Ib, beta subunit 30 kDa (PAFAH1B2), Synovial sarcoma translocation, chromosome 18 (SS18) and peroxisome biogenesis factor 1 (PEX1) were the most up-regulated. Moreover, Washizuka et al. (2009) showed that valproate, but not lithium, significantly increased the expression of the gene encoding for a subunit of mitochondrial complex I (NDUFV2) in LCLs from Japanese BD patients. In regard to other psychiatric phenotypes, unpublished data from LCLs of BD patients characterized for different risk of suicidal behaviour are showing that in vitro lithium treatment significantly perturbed the expression of the gene coding for the rate limiting enzyme spermidine/spermine N(1)-acethyltransferase (SAT1) (Squassina et al., in preparation).

Besides gene expression studies, LCLs have also been used to investigate the effect of lithium on protein levels in BD subjects. The study from Tseng et al. (2008) revealed that basal BDNF protein levels are decreased in LCLs from lithium responsive BD patients when compared with both their unaffected relatives and with healthy control participants. Interestingly, in vitro treatment with lithium of the LCLs decreased BDNF levels in all participants, but the difference between BD patients and healthy controls remained.

In addition, the pleiotropic effect of lithium on gene and protein expression has been deeply investigated in a series studies using animal (Bosetti et al., 2002; McQuillin et al., 2007; Chetcuti et al., 2008; Chen et al., 1999) and human (Sun et al., 2007; Seelan et al., 2008) cell tissues.

Specifically: 1) Lithium has been shown to increase the expression of the anti-apoptotic gene BCL2 with reduction of the expression of the pro-apoptotic genes p53 and Bax (Chen et al., 1999) clearly indicating a role in influencing the molecular cascade regulating the programmed cell death. This evidence acquires particularly interest in light of recent findings on BCL2. Two recent studies (Machado-Vieira et al., 2011, Uemura et al., 2011) demonstrated that, in individuals with BD, BCL2 gene expression regulated by the single nucleotide polymorphism (SNP) rs956572 directly impacted intracellular Ca2+ homeostasis dysregulation, a molecular signalling pathway proved to play a significant role in the pathogenesis of BD. 2) Using a genome wide gene expression approach (GWGE) on multiple prostate human cancer cell lines that were incubated with lithium, Sun and coworkers 11 showed a marked downregulation of genes involved in DNA replication. In another study, Seelan et al. (2008), in the attempt of profiling the lithium-modulated gene expression in human neuronal cells with microarray, identified peroxiredoxin 2 (PRDX2), an antioxidant enzyme, as the most upregulated gene, and tribbles homolog 3 (TRB3), a pro apoptotic protein, as the most downregulated, further suggesting a role of these pathways in the mood stabilization process.

In summary, lithium has been proven to significantly modulate the magnitude of the expression of a number of genes, among which the most robust and replicated changes were for BCL2, BAX, p53, and SAT1. Thus, we can take advantage of the well-established property of lithium of regulating the expression of these genes, and proteins, in a significant and stable manner. Conversely, these genes could be used as markers of the effect on lithium on the gene expression, providing a measure for the investigation of the effectiveness of EBV immortalization and repeated passages in eliminating the in vivo treatment effects.

Trial Objectives

This proposal aims to validate the assumption that LCLs, via EBV immortalization and repeated passages, are not influenced by environmental conditions, and especially drug treatment, at the time of sampling.

To do so, fresh lymphocytes and LCLs will be sampled in 20 healthy volunteers before (T0) and after (T1) four weeks of lithium treatment at a stable dose.

First, a set of molecular studies in fresh lymphocytes will examine the expression levels in target genes (namely BCL2, BAX, p53, SAT1) and protein (BDNF), and the activity of Complex I (all biological measures already known to be up-/down- regulated by lithium) at T0 and T1. These biological measures will serve as an assay sensitivity. We expect them to be regulated by in vivo lithium treatment and consequently to be significantly different between T0 and T1 in fresh lymphocytes.

Only the biological measures showing significant difference in fresh lymphocytes (not transformed with EBV) will be then analyzed in LCLs. Differential expression between LCLs sampled at T0 and T1 will indicate that the EBV transformation and repeated passages do not eliminate the environmental influences and, specifically, the effect of lithium treatment at sampling.

Finally, by studying healthy volunteers, we expect to decrease the confounding factors given by the presence of illness status.

ELIGIBILITY:
Inclusion Criteria:

* Men, ages 18 to 45 who are physically and mentally healthy.

Exclusion Criteria:

* Personal history of Axis I psychiatric disorders. Subjects with past, but not current (for at least 12 months) history of substance abuse will be eligible.
* Any medical conditions that represent contraindication to lithium use (for instance kidney or thyroid disease) and/or can potentially affect the gene expression profiles of the subjects.
* Ongoing treatment with drugs that have the potential of adverse interaction with lithium, for instance chronic use of NSAIDs, or diuretics.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05-05 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Expression levels of genes (known to be regulated by lithium) analyzed in lymphoblastoid cell cultures established from lymphocytes sampled in healthy volunteers before and after one month of lithium treatment. | 28 days
Expression levels of a protein, BDNF (known to be regulated by lithium) analyzed in lymphoblastoid cell cultures established from lymphocytes sampled in healthy volunteers before and after one month of lithium treatment. | 28 days
Enzymatic activity of Complex I (known to be altered by lithium) analyzed in lymphoblastoid cell cultures established from lymphocytes sampled in healthy volunteers before and after one month of lithium treatment. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin Alda, MD, FRCPC, Study Chair — Dalhousie University
Locations (1):
- Department of Psychiatry, Abbie J Lane Building, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Baldessarini RJ, Tondo L. Does lithium treatment still work? Evidence of stable responses over three decades. Arch Gen Psychiatry. 2000 Feb;57(2):187-90. doi: 10.1001/archpsyc.57.2.187. PMID 10665622
- [Background] Garnham J, Munro A, Slaney C, Macdougall M, Passmore M, Duffy A, O'Donovan C, Teehan A, Alda M. Prophylactic treatment response in bipolar disorder: results of a naturalistic observation study. J Affect Disord. 2007 Dec;104(1-3):185-90. doi: 10.1016/j.jad.2007.03.003. Epub 2007 Apr 17. PMID 17442400
- [Background] Sun X, Young LT, Wang JF, Grof P, Turecki G, Rouleau GA, Alda M. Identification of lithium-regulated genes in cultured lymphoblasts of lithium responsive subjects with bipolar disorder. Neuropsychopharmacology. 2004 Apr;29(4):799-804. doi: 10.1038/sj.npp.1300383. PMID 14735134
- [Background] Sugawara H, Iwamoto K, Bundo M, Ishiwata M, Ueda J, Kakiuchi C, Ishigooka J, Kato T. Effect of mood stabilizers on gene expression in lymphoblastoid cells. J Neural Transm (Vienna). 2010 Feb;117(2):155-64. doi: 10.1007/s00702-009-0340-8. Epub 2009 Dec 1. PMID 19949822
- [Background] Washizuka S, Iwamoto K, Kakiuchi C, Bundo M, Kato T. Expression of mitochondrial complex I subunit gene NDUFV2 in the lymphoblastoid cells derived from patients with bipolar disorder and schizophrenia. Neurosci Res. 2009 Mar;63(3):199-204. doi: 10.1016/j.neures.2008.12.004. Epub 2008 Dec 24. PMID 19135101
- [Background] Tseng M, Alda M, Xu L, Sun X, Wang JF, Grof P, Turecki G, Rouleau G, Young LT. BDNF protein levels are decreased in transformed lymphoblasts from lithium-responsive patients with bipolar disorder. J Psychiatry Neurosci. 2008 Sep;33(5):449-53. PMID 18787660
- [Background] Bosetti F, Seemann R, Bell JM, Zahorchak R, Friedman E, Rapoport SI, Manickam P. Analysis of gene expression with cDNA microarrays in rat brain after 7 and 42 days of oral lithium administration. Brain Res Bull. 2002 Jan 15;57(2):205-9. doi: 10.1016/s0361-9230(01)00744-4. PMID 11849827
- [Background] McQuillin A, Rizig M, Gurling HM. A microarray gene expression study of the molecular pharmacology of lithium carbonate on mouse brain mRNA to understand the neurobiology of mood stabilization and treatment of bipolar affective disorder. Pharmacogenet Genomics. 2007 Aug;17(8):605-17. doi: 10.1097/FPC.0b013e328011b5b2. PMID 17622937
- [Background] Chetcuti A, Adams LJ, Mitchell PB, Schofield PR. Microarray gene expression profiling of mouse brain mRNA in a model of lithium treatment. Psychiatr Genet. 2008 Apr;18(2):64-72. doi: 10.1097/YPG.0b013e3282fb0051. PMID 18349697
- [Background] Chen RW, Chuang DM. Long term lithium treatment suppresses p53 and Bax expression but increases Bcl-2 expression. A prominent role in neuroprotection against excitotoxicity. J Biol Chem. 1999 Mar 5;274(10):6039-42. doi: 10.1074/jbc.274.10.6039. PMID 10037682
- [Background] Sun A, Shanmugam I, Song J, Terranova PF, Thrasher JB, Li B. Lithium suppresses cell proliferation by interrupting E2F-DNA interaction and subsequently reducing S-phase gene expression in prostate cancer. Prostate. 2007 Jun 15;67(9):976-88. doi: 10.1002/pros.20586. PMID 17440966
- [Background] Seelan RS, Khalyfa A, Lakshmanan J, Casanova MF, Parthasarathy RN. Deciphering the lithium transcriptome: microarray profiling of lithium-modulated gene expression in human neuronal cells. Neuroscience. 2008 Feb 19;151(4):1184-97. doi: 10.1016/j.neuroscience.2007.10.045. Epub 2007 Nov 13. PMID 18222042
- [Background] Machado-Vieira R, Pivovarova NB, Stanika RI, Yuan P, Wang Y, Zhou R, Zarate CA Jr, Drevets WC, Brantner CA, Baum A, Laje G, McMahon FJ, Chen G, Du J, Manji HK, Andrews SB. The Bcl-2 gene polymorphism rs956572AA increases inositol 1,4,5-trisphosphate receptor-mediated endoplasmic reticulum calcium release in subjects with bipolar disorder. Biol Psychiatry. 2011 Feb 15;69(4):344-52. doi: 10.1016/j.biopsych.2010.10.019. Epub 2010 Dec 16. PMID 21167476
- [Background] Uemura T, Green M, Corson TW, Perova T, Li PP, Warsh JJ. Bcl-2 SNP rs956572 associates with disrupted intracellular calcium homeostasis in bipolar I disorder. Bipolar Disord. 2011 Feb;13(1):41-51. doi: 10.1111/j.1399-5618.2011.00897.x. PMID 21320251